CLINICAL TRIAL: NCT00452816
Title: Marketing Workplace Chronic Disease Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); American Cancer Society, Inc. (Other)
Responsible Party: Jeffrey Harris, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-4829-E/G 01; CDC Grant 1 PO1 CD000249-01
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Health Behavior; Chronic Disease
Keywords: Chronic Disease; Employer Health Costs; Health Promotion; Insurance Benefits; Marketing of Health Services; Mass Screening; Prevention & Control; Tobacco Use Cessation; Workplace
MeSH Terms: conditions — Health Behavior; Chronic Disease; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intervention Group - Workplace Solutions Consulting
  Interventions: Behavioral: Workplace Solutions Consulting approach
- 2 (Active Comparator): Delayed Intervention
  Interventions: Behavioral: Delayed intervention

INTERVENTIONS:
Behavioral: Workplace Solutions Consulting approach — Consulting process includes:
  1. baseline measure of best practices
  2. gap analysis and recommendations reporting
  3. delivery of "solution set" toolkits for each practice chosen for implementation
  Arms: Intervention
Behavioral: Delayed intervention — Abbreviated version of the Workplace Solutions Consulting process applied in the intervention group
  Arms: 2

SUMMARY:
The objective of the project is to understand how best to help mid-size employers adopt evidence-based chronic disease prevention practices that improve employee health behaviors.

DETAILED DESCRIPTION:
Employers have the incentive and the means to play a key role in chronic disease prevention. The incentive - employers need to control the costly and growing burden of chronic diseases among their employees. The means - employers purchase 94% of private health insurance, and employees spend one third of their lives in the workplace, where they often eat, move, socialize, and smoke. Over the past 5 years, the CDC and the Task Force on Community Preventive Services have recommended a number of chronic disease prevention practices. Among these, we have identified 17 practices that employers should adopt. These practices include health insurance benefits, workplace policies, and workplace programs, and aim at increasing employees' disease screening, healthy eating, influenza immunization, physical activity and tobacco cessation. Unfortunately, employer surveys reveal low adoption of these practices.

Working with the American Cancer Society, our research team from the University of Washington has developed and pilot-tested an innovative consulting intervention to increase adoption of these practices. Our two-stage intervention is comprehensive yet tailored by employer feedback.

The intervention:

* markets the "business case" that employers can help control health-care costs and productivity losses through adoption of these practices
* enables implementation by providing tools for each practice.

In this proposal, our primary aim is to test this intervention in a randomized, controlled trial among 48 medium-sized employers with a high proportion of socioeconomically disadvantaged employees in the Puget Sound area. Our primary outcome is change in employer practices as measured by survey and validated by audit and contract and policy review.

Our secondary aims include:

* development and pilot-testing of an employee-level health risk behavior survey
* cost analysis and assessment of feasibility of our intervention
* assessment of employees' preference for different message sources and message appeals.

Our multidisciplinary research team includes business, communication, and public health faculty and has more than 10 years of experience in both chronic disease prevention and working with business. If successful, our team's approach has broad applicability to other public health problems.

ELIGIBILITY:
Inclusion Criteria:

* Corporate size equal to 100 to 999 part-time and full-time employees (excluding seasonal and temporary workers)
* Headquarters located in King County, Washington, and in a zip code within a 30 mile radius of the research center
* Within an industry with an average annual salary below the median annual salary for King County, Washington (defined by 3-digit NAICS code)
* 50% or more employees are age 35 or older

Exclusion Criteria:

* Do not offer health insurance to full-time employees
* In existence for less than 3 years
* No physical address to which employees report
* Current or previous participation in other workplace health promotion study
* Recent refuser or non-responder for other current workplace health promotion study
* Current participant in other American Cancer Society employer program
* Not willing to be randomized to intervention or comparison group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in employer practices in health benefits, policies and programs | 15 month follow-up survey

SECONDARY OUTCOMES:
Development and pilot-testing of an employee-level health risk behavior survey | within 12 months of recruitment completion
Cost analysis and assessment of feasibility of this intervention | within 15 months of recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Harris, MD, MPH, MBA, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Hannon PA, Harris JR, Sopher CJ, Kuniyuki A, Ghosh DL, Henderson S, Martin DP, Weaver MR, Williams B, Albano DL, Meischke H, Diehr P, Lichiello P, Hammerback KE, Parks MR, Forehand M. Improving low-wage, midsized employers' health promotion practices: a randomized controlled trial. Am J Prev Med. 2012 Aug;43(2):125-33. doi: 10.1016/j.amepre.2012.04.014. PMID 22813676